CLINICAL TRIAL: NCT00998608
Title: A Randomized, Double-Blind, Comparison of the Efficacy and Safety of Risperidone Versus Risperidone Combined With Low Dose of Haloperidol in the Treatment of Schizophrenic Disorder
Brief Title: Comparison of the Efficacy and Safety of Risperidone Versus Risperidone Plus Low Dose of Haloperidol in the Treatment of Schizophrenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated
Sponsor: Kaohsiung Kai-Suan Psychiatric Hospital (Other Government)
Responsible Party: Ching-Hua Lin, M.D., Kaohsiung Kai-Suan Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KSPH-2007-17
Record Dates: First submitted 2009-10-08; First posted 2009-10-20 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HR (Experimental): risperidone 2mg/d + haloperidol 2mg/d
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: risperidone — risperidone 4mg/d

SUMMARY:
The purpose of this study is to compare the efficacy and safety of risperidone and risperidone plus low dose of haloperidol in the acutely schizophrenic patients.

DETAILED DESCRIPTION:
Antipsychotic monotherapy is recognized as the treatment of choice for patients with schizophrenia. Surveys have shown that antipsychotic drug combinations are frequently prescribed, yet few clinical studies have examined this practice. Risperidone, an atypical antipsychotics, has low incidence of extrapyramidal symptom (EPS) but with high cost compared to haloperidol. It has been reported that a relatively low daily dose of haloperidol at which individual patients develop slightly increase in EPS and has neurocognitive benefits as risperidone. The objective of the study is to compare the efficacy and safety of the fixed-dosed risperidone and risperidone combined with haloperidol in the treatment of acute psychotic exacerbations of schizophrenia.In this 6-week, double-blind, fixed-dose study, patients with schizophrenic disorder (DSM-IV diagnosis) are randomly assigned to risperidone (4 mg/d) or risperidone (2 mg/d) plus haloperidol (2 mg/d). The hypothesis is that the two treatment groups have the similar efficacy and safety, but different cost. The primary efficacy measure is change from baseline in Positive and Negative Syndrome Scale (PANSS) total scores; secondary outcomes include Clinical Global Impression-Change (CGI-C), the Calgary Depression Scale for Schizophrenics (CDSS), subject-reported outcomes via the Short Form-36 (SF-36), auditory evoked potentials (AEPs), and cognitive and social functioning. Safety assessments include the change from baseline on Simpson-Angus Rating Scale (SAS), Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Scale (BAS), and UKU Side-effects Rating Scale (UKU), and the change from baseline in prolactin levels, body weight, AC glucose level, lipid panel (cholesterol, high density lipid protein [HDL], low density lipid protein [LDL], and triglyceride [TG])

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Clinical Global Impression large than 3
* Written informed consent

Exclusion Criteria:

* Comorbid of substance abuse/dependence
* Present or history of tardive dyskinesis or neuroleptic malignant syndromes
* Severe physical problems
* pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
change from baseline in Positive and Negative Syndrome Scale (PANSS) total scores | 6 weeks after the initiation of antipsychotic use

CONTACTS AND LOCATIONS:
Overall Officials: Li-Shiu Chou, M.D., Study Director — Kai-Suan Psychiatric Hospital
Locations (1):
- Kai-Suan Psychiatric Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Result] Tapp A, Wood AE, Secrest L, Erdmann J, Cubberley L, Kilzieh N. Combination antipsychotic therapy in clinical practice. Psychiatr Serv. 2003 Jan;54(1):55-9. doi: 10.1176/appi.ps.54.1.55. PMID 12509667
- [Result] Centorrino F, Goren JL, Hennen J, Salvatore P, Kelleher JP, Baldessarini RJ. Multiple versus single antipsychotic agents for hospitalized psychiatric patients: case-control study of risks versus benefits. Am J Psychiatry. 2004 Apr;161(4):700-6. doi: 10.1176/appi.ajp.161.4.700. PMID 15056517
- [Result] Lehman AF, Lieberman JA, Dixon LB, McGlashan TH, Miller AL, Perkins DO, Kreyenbuhl J; American Psychiatric Association; Steering Committee on Practice Guidelines. Practice guideline for the treatment of patients with schizophrenia, second edition. Am J Psychiatry. 2004 Feb;161(2 Suppl):1-56. No abstract available. PMID 15000267
- [Result] Woods SW. Chlorpromazine equivalent doses for the newer atypical antipsychotics. J Clin Psychiatry. 2003 Jun;64(6):663-7. doi: 10.4088/jcp.v64n0607. PMID 12823080
- [Result] McEvoy JP, Hogarty GE, Steingard S. Optimal dose of neuroleptic in acute schizophrenia. A controlled study of the neuroleptic threshold and higher haloperidol dose. Arch Gen Psychiatry. 1991 Aug;48(8):739-45. doi: 10.1001/archpsyc.1991.01810320063009. PMID 1883257